CLINICAL TRIAL: NCT02210000
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Effect of 12 Weeks of Once-daily Dosing of the Oral Motilin Receptor Agonist Camicinal, on Gastroparesis Symptoms in Type 1 and 2 Diabetic Subjects With Gastroparesis
Brief Title: A Study to Evaluate the Effect of Camicinal on Gastroparesis Symptoms in Type 1 and 2 Diabetic Subjects With Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201159
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-09

CONDITIONS: Gastroparesis
Keywords: repeat dose; phase II; GCSI-DD; pharmacodynamics; gastroparesis; type 1 and type 2 diabetes mellitus; camicinal; GSK962040; symptoms; gut motility
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus, Type 2 | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive camicinal matching placebo orally once daily (QD) from Day 1 to Day 84
  Interventions: Drug: Placebo
- Camicinal 25mg (Experimental): Subjects will receive camicinal 25 mg orally QD from Day 1 to Day 84
  Interventions: Drug: Camicinal

INTERVENTIONS:
Drug: Placebo — Camicinal matching placebo is available as tablet to be taken orally with 100mL of water in the morning
  Arms: Placebo
Drug: Camicinal — Camicinal is available as 25 mg tablet to be taken orally with 100mL of water in the morning
  Arms: Camicinal 25mg

SUMMARY:
This study is a randomized, double-blind, placebo controlled trial designed to confirm the symptomatic effects of camicinal treatment vs. placebo, on gastroparesis symptoms in type 1 and 2 diabetic subjects with gastroparesis. The primary purpose of this study is to determine if a low-dose of camicinal (25 milligram[mg]) for 12 weeks of repeat administration improves gastroparesis symptoms as measured by the Gastrointestinal Cardinal Symptom Index - Daily Diary (GCSI-DD) in approximately 120 subjects with type 1 or 2 diabetes mellitus (DM) who have documented abnormally slow gastric emptying and have symptoms consistent with gastroparesis.

Subjects will be randomized in a 1:1 ratio to receive either camicinal or placebo. The study will consist of a screening/baseline period of up to 35 days, a 12 week treatment period, a 2-week post-treatment assessment of symptoms and a 14 day (+/- 2 days) post treatment safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes mellitus (acetylated hemoglobin A1 [HbA1c] <=11.0%)
* Male or female between 18 and 80 years of age, inclusive.
* Patient has gastroparesis at screening. A patient is eligible if one of the following criteria are met: Gastric half-time of emptying >upper limit of normal as determined by Carbon-13 radioisotope (C13) oral breath test; % C13-dose recovered < lower limit of normal at 90 or 120 minutes
* Patient must report a >=3 month history of relevant symptoms of gastroparesis (e.g., chronic post-prandial fullness, early satiety, post-prandial nausea).
* Patients will have a mean of the daily scores over a minimum of 7 days indicating >= mild (2) severity for the fullness/early satiety subscale as assessed using the GCSI-DD during the screening period prior to randomization.
* A female patient is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 milli international units per milliliter [mIU/mL], or a value consistent with the local laboratory standard value, is confirmatory) or is of child-bearing potential and agrees to use contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female patients must agree to use contraception for at least 5 days following the last dose of study medication.
* Body mass index (BMI) >18 and <=42.0 kilogram per meter square (kg/m^2) (inclusive).
* QTc <450 millisecond (msec) or QTc <480 msec in patients with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period. The QT correction formula (Bazett's, Fridericia's, etc) used to determine inclusion and discontinuation should be the same throughout the study.
* Aspartate aminotransferase and alanine aminotransferase <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Patient has acute severe gastroenteritis
* Patient has a gastric pacemaker
* Patient is on chronic enteral (e.g., feeding tube) or parenteral feeding
* Recent (last 6 weeks) history of poor control of diabetes e.g. hypoglycaemia requiring medical intervention, diabetic ketoacidosis, admission for control of diabetes or complications of diabetes
* Patient has evidence of severe cardiovascular autonomic neuropathy (e.g. history of recurrent syncope in the last 6 months)
* Patient has a history of eating disorders (anorexia nervosa, binge eating, bulimia)
* Use of medications potentially influencing upper gastrointestinal motility or appetite at least 1 week prior to screening (e.g., prokinetic drugs, macrolide antibiotics [erythromycin], glucagon-like peptide-1 [GLP-1] mimetics)
* Patient has had intrapyloric botox injections.
* A patient would be eligible if the botox treatment was in the past (>6 months previously) and was not being repeated.
* Patient has had a gastrectomy, or major gastric surgical procedure or any evidence of bowel obstruction or strictures within the previous 12 months
* Dosage of any concomitant medications has not been stable for at least 3 weeks, except for routine adjustments in daily insulin treatments.
* Estimated (or measured) glomerular filtration rate <=30 mL/minute.
* Daily opiate use at screening
* Use of prohibited medications that potentially influence upper gastrointestinal motility or appetite, or medications that may interfere with the methods of measuring gastric emptying e.g., prokinetic drugs, macrolide antibiotics (erythromycin, azithromycin), GLP-1 mimetics, anti-cholinergics, chronic/regular use of opiates
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease (including liver disease or known hepatic or biliary abnormalities, with the exception of Gilbert's syndrome or asymptomatic gallstones) or other condition that would in the opinion of the investigator or medical monitor make the subject unsuitable for inclusion in this clinical study.
* Concurrent enrollment in any other interventional study/(ies) involving a novel (i.e. unapproved or experimental) chemical or biopharmaceutical entity.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline Medical Monitor, contraindicates their participation.
* Lactating or Pregnant females as determined by positive serum or urine human chorionic gonadotropin test (from the first urine of the day) at screening or prior to dosing.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2015-08-24 (Actual); Study Completion 2015-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (32):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Wyoming, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Mentor, Ohio
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Spring, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 27 August 2014 till 24 August 2015 across 34 centers in the united states (US). A total of 120 participants with gastroparesis and Type 1 or 2 diabetes mellitus were planned to be enrolled.
Pre-assignment Details: A total of 387 participants with gastroparesis and Type 1 or 2 diabetes mellitus were screened, of which 273 participants did not meet the inclusion/exclusion criteria and thus, were screen failures. A total of 114 participants were randomized in the study. Participants started recording GCSI-DD for 7 days post-screening to assess baseline symptoms
Groups:
- CAMICINAL 25 MG: Eligible participants received oral Camicinal 25 milligrams (mg) once daily in the morning with 100 milliliter (mL) of water up to 84 days and were followed-up for 2 weeks.
- PLACEBO: Eligible participants received oral matching Placebo once daily in the morning with 100 mL of water up to 84 days and were followed-up for 2 weeks.
Period: Overall Study
Arm/Group | CAMICINAL 25 MG | PLACEBO
Started | 57 | 57
Completed | 38 | 36
Not Completed | 19 | 21
Not completed — Study Terminated | 11 | 12
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least one dose of the study drug and were followed-up for at least one post-baseline safety assessment; however, one participant randomized to Placebo arm had quantifiable concentration of camicinal in blood and therefore was analyzed in the camicinal group.
Groups:
- CAMICINAL 25 MG: Eligible participants received oral Camicinal 25 mg once daily in the morning with 100 mL of water up to 84 days and were followed-up for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | CAMICINAL 25 MG | PLACEBO | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (12.47) | 58.3 (9.81) | 57.8 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 42 | 36 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 44 | 40 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Based on the Fullness/Early Satiety Subscale (Responders) as Assessed by Gastrointestinal Cardinal Symptom Index-Daily Diary (GCSI-DD) at Week 12
Description: The GCSI-DD consists of nine symptom severity items covering the following domains: nausea/vomiting; fullness/early satiety, and bloating. In addition, the GCSI-DD contains two symptom severity items upper abdominal pain and overall rating of gastroparesis symptoms. Participants were asked to rate each symptom on a 6-point scale from 0 to 5 with lower scores representing less symptom severity and higher scores indicating more severe symptoms. Fullness/early satiety response is defined as an improvement from Baseline by at least one point in the weekly average for the subscale. A participant was defined as a responder if the participant's weekly average change from Baseline in the fullness/early satiety response score improved by at least 1 point. Percentage of participants showing response were presented.
Time Frame: Week 12
Population: Intent-to-treat (ITT) Population comprised of all randomized participants.
Measure: Number; unit: Percentage of responders
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 57 | 57
Percentage of responders | 26.32 | 42.11
Statistical Analysis 1: Comparison: CAMICINAL 25 MG vs PLACEBO; Test type: Superiority; p = 0.017, Bayesian method — Posterior probability of the treatment difference in response rate at Week 12 being greater than 0%; Median Difference (Net) = -0.212, 95% CI 2-sided [-0.3716 to -0.0448]

2. Secondary Outcome: Change From Baseline in Individual Items, Subscales and Total Score of GCSI-DD at Week 12
Description: Items of GCSI-DD for gastroparesis (GP) symptom assessment included: 3-nausea, 4-feeling full after meals, 5-bloating, 6-unable to finish normal meal, 7-retching, 8-vomiting, 9-stomach visibly larger, 10-stomach fullness, 11-loss of appetite, 12-upper abdominal pain, 13-upper abdominal discomfort and 14-overall severity of GP symptoms. Each symptom rated on a 6-point scale from 0 to 5 where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Score of nausea/vomiting subscale was mean of items 3, 7, 8; fullness/early satiety subscale was mean of items 4, 6, 10, 11; bloating subscale was mean of items 5, 9. Total GCSI-DD score was mean of 3 subscales. For all, 0 indicated absence of symptom and higher score indicated greater severity of symptoms. Baseline was defined as weekly average of last 7 daily scores recorded during screening period. Change from Baseline was calculated by subtracting mean score for Baseline from weekly average score of Week 12.
Time Frame: Baseline (Screening) and Week 12
Population: ITT Population. Only those participants available at the time of assessment were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 57 | 57
Scores on a scale
  Nausea: number analyzed (Participants) | 34 | 32
  Nausea | -1.250 (0.1714) | -1.460 (0.1765)
  Feeling full after meals: number analyzed (Participants) | 34 | 32
  Feeling full after meals | -1.063 (0.2102) | -1.812 (0.2146)
  Bloating: number analyzed (Participants) | 34 | 32
  Bloating | -1.382 (0.2227) | -1.871 (0.2270)
  Unable to finish normal meal: number analyzed (Participants) | 34 | 32
  Unable to finish normal meal | -0.876 (0.1819) | -1.373 (0.1858)
  Retching: number analyzed (Participants) | 34 | 32
  Retching | -0.894 (0.1517) | -0.944 (0.1554)
  Vomiting: number analyzed (Participants) | 34 | 32
  Vomiting | -0.532 (0.1112) | -0.494 (0.1144)
  Stomach visiblly larger: number analyzed (Participants) | 34 | 32
  Stomach visiblly larger | -0.998 (0.2124) | -1.473 (0.2165)
  Stomach fullness: number analyzed (Participants) | 34 | 32
  Stomach fullness | -1.200 (0.2090) | -1.661 (0.2124)
  Loss of appetite: number analyzed (Participants) | 34 | 32
  Loss of appetite | -0.930 (0.1732) | -1.465 (0.1774)
  Upper abdominal pain | -1.186 (0.1887) | -1.383 (0.1922)
  Upper abdominal discomfort: number analyzed (Participants) | 34 | 32
  Upper abdominal discomfort | -1.304 (0.2051) | -1.618 (0.2097)
  Overall severity of GP: number analyzed (Participants) | 34 | 32
  Overall severity of GP | -1.173 (0.1626) | -1.557 (0.1667)
  Nausea/vomiting subscale: number analyzed (Participants) | 34 | 32
  Nausea/vomiting subscale | -0.888 (0.1183) | -0.956 (0.1216)
  Fullness/Early Satiety Subscale: number analyzed (Participants) | 34 | 32
  Fullness/Early Satiety Subscale | -1.041 (0.1696) | -1.589 (0.1725)
  Bloating Subscale | -1.189 (0.2115) | -1.668 (0.2153)
  Total GCSI-DD scale | -1.037 (0.1470) | -1.393 (0.1498)
Statistical Analysis 1: Comparison: CAMICINAL 25 MG vs PLACEBO; Nausea at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.210, 95% CI 2-sided [-0.2353 to 0.6553] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 2: Comparison: CAMICINAL 25 MG vs PLACEBO; Feeling full after meals at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.749, 95% CI 2-sided [0.2275 to 1.2705] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 3: Comparison: CAMICINAL 25 MG vs PLACEBO; Bloating at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.489, 95% CI 2-sided [-0.0592 to 1.0374] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 4: Comparison: CAMICINAL 25 MG vs PLACEBO; Not able to finish meal at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.497, 95% CI 2-sided [0.0396 to 0.9550] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 5: Comparison: CAMICINAL 25 MG vs PLACEBO; Retching at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.3386 to 0.4395] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 6: Comparison: CAMICINAL 25 MG vs PLACEBO; Vomiting at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = -0.038, 95% CI 2-sided [-0.3242 to 0.2492] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 7: Comparison: CAMICINAL 25 MG vs PLACEBO; Stomach visibly larger at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.475, 95% CI 2-sided [-0.0483 to 0.9978] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 8: Comparison: CAMICINAL 25 MG vs PLACEBO; Stomach fullness at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.461, 95% CI 2-sided [-0.0519 to 0.9748] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 9: Comparison: CAMICINAL 25 MG vs PLACEBO; Loss of appetite at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.536, 95% CI 2-sided [0.0967 to 0.9745] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 10: Comparison: CAMICINAL 25 MG vs PLACEBO; Upper abdominal pain at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.196, 95% CI 2-sided [-0.2746 to 0.6671] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 11: Comparison: CAMICINAL 25 MG vs PLACEBO; Upper abdominal discomfort at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.314, 95% CI 2-sided [-0.2013 to 0.8292] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 12: Comparison: CAMICINAL 25 MG vs PLACEBO; Overall severity of your GP symptoms at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.384, 95% CI 2-sided [-0.0323 to 0.7997] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 13: Comparison: CAMICINAL 25 MG vs PLACEBO; Nausea/Vomiting Subscale at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.068, 95% CI 2-sided [-0.2366 to 0.3723] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 14: Comparison: CAMICINAL 25 MG vs PLACEBO; Fullness/Early Satiety Subscale at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.548, 95% CI 2-sided [0.1333 to 0.9628] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 15: Comparison: CAMICINAL 25 MG vs PLACEBO; Bloating Subscale at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.479, 95% CI 2-sided [-0.0386 to 0.9966] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo
Statistical Analysis 16: Comparison: CAMICINAL 25 MG vs PLACEBO; Total GCSI-DD at Week 12. The least square means were the adjusted means which had been estimated with a mixed model using Baseline weekly average value, diabetes type, treatment, week and the interaction between treatment and week as fixed effects, participants as random effect and week as repeated effect; Test type: Superiority; Mean Difference (Net) = 0.356, 95% CI 2-sided [-0.0049 to 0.7179] — A negative difference indicated greater improvement in the Camicinal group compared to Placebo

3. Secondary Outcome: Number of Participants With Change From Baseline (Day 1) in Blood Pressure of Potential Clinical Importance (PCI) Over 100 Days
Description: Abnormal values of systolic and diastolic blood pressure were measured. If the value for a participant at a given visit was outside the PCI, the participants were further categorized as per the increase or decrease of systolic blood pressure (SBP) and diastolic blood pressure (DBP) from Baseline by 10, 20 and 40 millimeters of mercury (mm of Hg). Number of participants with absolute (ABS) SBP (>160 mm Hg) and ABS DBP (100 mm Hg) were also analyzed. Change from Baseline (CFB) is the post-Baseline value minus the Baseline value. Participants were counted only once per parameter. Participant may have had more than 1 abnormal parameter. Only worst post-Baseline CFB values were considered. The categories mentioned for data values indicate the blood pressure ranges of clinical concern.
Time Frame: Up to 100 days
Population: Safety Population comprised of participants who received at least one dose of the study drug and were followed-up for at least one post-Baseline safety assessment; however, one participant randomized to Placebo arm had quantifiable concentration of Camicinal in blood and therefore was analyzed in the Camicinal group.
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  SBP, ABS: > 160 | 4 | 5
  SBP, CFB: INCREASE >=20 | 12 | 7
  SBP, CFB: INCREASE >=40 | 1 | 2
  SBP, CFB: DECREASE >=20 | 9 | 11
  SBP, CFB: DECREASE >=40 | 0 | 2
  DBP, ABS: >100 | 1 | 2
  DBP, CFB: INCREASE >=10 | 13 | 10
  DBP, CFB: INCREASE >=20 | 1 | 1
  DBP, CFB: DECREASE >=20 | 8 | 19
  DBP, CFB: DECREASE >=10 | 3 | 2

4. Secondary Outcome: Number of Participants With Change From Baseline (Day 1) in Heart Rate of PCI Over 100 Day
Description: Abnormal values of heart rate over 100 days was analyzed and reported. Participants were counted only once per parameter. Participant may have had more than 1 abnormal parameter. Only worst post baseline CFB values were considered. The categories mentioned for data values indicate the heart rate ranges of clinical concern.
Time Frame: Up to 100 days
Population: Safety Population. One participant randomized to Placebo arm had quantifiable concentration of Camicinal in blood and therefore was analyzed in the Camicinal group.
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  ABS: >110 | 1 | 1
  CFB: INCREASE >=15 | 4 | 4
  CFB: INCREASE >=30 | 0 | 2
  CFB: DECREASE >=15 | 5 | 7
  CFB: DECREASE >=30 | 1 | 0

5. Secondary Outcome: Number of Participants With Normal and Abnormal 12-lead Electrocardiogram (ECG) Measurements Over 100 Days
Description: The 12-lead ECG was analyzed as a measure of safety and tolerability. Number of participants with normal ECG, abnormal clinically significant, and abnormal clinically not significant ECG were reported. PR interval of < 110 and > 220 milliseconds (msec), QRS interval of <75 and > 110 msec, absolute QTc interval of > 450 to ≤ 480 or > 480 to ≤ 500 or >500 msec, and increase from Baseline in QTc of > 30 to ≤ 60 msec or >60 msec was considered as of abnormal.
Time Frame: Up to 100 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  BASELINE, NORMAL | 34 | 29
  BASELINE, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 24 | 26
  BASELINE, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 1
  DAY 14, NORMAL | 32 | 25
  DAY 14, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 22 | 25
  DAY 14, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 0
  DAY 28, NORMAL | 24 | 22
  DAY 28, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 28 | 24
  DAY 28, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 0
  DAY 56, NORMAL | 19 | 23
  DAY 56, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 25 | 19
  DAY 56, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 0
  DAY 84, NORMAL | 18 | 21
  DAY 84, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 20 | 15
  DAY 84, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 0
  FOLLOW-UP, NORMAL | 32 | 28
  FOLLOW-UP, ABNORMAL - NOT CLINICALLY SIGNIFICANT | 24 | 25
  FOLLOW-UP, ABNORMAL - CLINICALLY SIGNIFICANT | 0 | 0

6. Secondary Outcome: Number of Participants With Change From Baseline in Hematological Abnormalities of PCI by Treatment and Visit Over Period
Description: Hematology analysis was performed at screening (fasted) and during the study at each indicated time point. Participants with abnormalities in changes from Baseline values were recorded. Total absolute neutrophil count (tANC <1.5 Giga per Liter [G/L]), hemoglobin (<25 or >25 G/L), hematocrit (<0.075 or >0.075 %), platelet count (<100 or >500 G/L), lymphocytes low (<0.8 G/L), and white blood cells (WBC <3 G/L or >20G/L) were analyzed for their low (L) or high (H) values. Change from Baseline (CFB) was the post-Baseline value minus then Baseline value. Baseline was defined as last non-missing measurement prior to dosing. One participant was randomized to Placebo arm; however, was included within the Camicinal treatment group as they reported at least one PK trough concentration >53 nano-grams per milliliter (ng/mL).
Time Frame: Up to 100 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  tANC, L, <1.5, Day 56 | 0 | 1
  tANC, L, <1.5, Day 100 | 0 | 1
  Hemoglobin, H, CFB >25, Day 56 | 1 | 0
  Hemoglobin, H, CFB >25, Day 84 | 1 | 0
  Hemoglobin, L, CFB < -25, Day 100 | 1 | 0
  Hemoglobin, H, CFB >25, Day 100 | 1 | 0
  Hematocrit, H, >0.54, Day 1 | 0 | 1
  Hematocrit, H, >0.54, Day 28 | 0 | 1
  Hematocrit, H, >0.54, Day 56 | 0 | 1
  Hematocrit, H, CFB >0.075, Day 56 | 1 | 0
  Hematocrit, H, CFB >0.075, Day 84 | 1 | 0
  Hematocrit, L, CFB, >0.54, Day 100 | 1 | 0
  Hematocrit, L, CFB, < -0.075, Day 100 | 1 | 0
  Hematocrit, H, CFB, >0.075, Day 100 | 1 | 0
  Platelet count, L, <100, Day 1 | 1 | 0
  Platelet count, L, <100, Day 28 | 1 | 0
  Platelet count, L, <100, Day 100 | 1 | 0
  Lymphocytes, L, <0.8, Day 1 | 1 | 0

7. Secondary Outcome: Number of Participants With Change From Baseline Clinical Chemistry Abnormalities of PCI by Treatment and Visit Over Period
Description: Clinical chemistry laboratory analysis was performed at screening (fasted) and during the study at each indicated time point. Albumin low (<30 G/L), calcium low (<2 or >2.75 millimoles per Liter [mmol/L]), creatinine (>44 micromoles per Liter change from baseline), Glucose (<3 or >18 mmol/L), potassium (<3.0 or >5.5 mmol/L), sodium (<130 or >150 mmol/L), and carbon di oxide (CO2) (<18 or >35 mmol/L) were analyzed for their low (L) or high (H) values. Participants with abnormalities in changes from Baseline values were recorded. Change from Baseline is the post-Baseline value minus the Baseline value.
Time Frame: Up to 100 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  Creatinine, H, CFB>44, Day 28 | 1 | 0
  Creatinine, H, CFB>44, Day 56 | 0 | 1
  Creatinine, H, CFB>44, Day 84 | 2 | 2
  Glucose, H, >18, Day 1 | 1 | 3
  Glucose, H, >18, Day 28 | 1 | 4
  Glucose, L, <3.0, Day 56 | 1 | 0
  Glucose, H, >18, Day 56 | 2 | 3
  Glucose, H, >18, Day 84 | 2 | 2
  Glucose, H, >18, Day 100 | 2 | 2
  Potassium, H, >5.5, Day 1 | 0 | 2
  Potassium, H, >5.5, Day 28 | 2 | 0
  Potassium, H, >5.5, Day 56 | 3 | 2
  Potassium, H, >5.5, Day 84 | 1 | 1
  Potassium, H, >5.5, Day 100 | 1 | 0
  Sodium, L, <130, Day 84 | 1 | 0
  Sodium, L, <130, Day 100 | 0 | 1
  Carbon di oxide, L, <18, Day 1 | 1 | 2
  Carbon di oxide, L, <18, Day 28 | 1 | 0
  Carbon di oxide, L, <18, Day 56 | 1 | 0
  Carbon di oxide, L, <18, Day 84 | 1 | 1
  Carbon di oxide, L, <18, Day 100 | 1 | 3

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs), and Adverse Events Leading to Discontinuation of the Study Drug
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above. Any AE or SAE that led discontinuation of the study drug either by participant or by investigator was considered as an AE leading to discontinuation of the study drug.
Time Frame: Up to end of follow up (100 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 56
Participants
  WITH ANY AE | 28 | 35
  WITH ANY SAE | 3 | 2
  WITH AE LEADING TO DISCONTINUATION | 2 | 5

9. Secondary Outcome: Trough Plasma Concentration of Camicinal on Day 28 and Day 84
Description: A pre-dose blood sample was collected on Days 28 and 84 for pharmacokinetic analysis. This analysis was applicable only for Camicinal arm and thus, no participants from Placebo arm were analyzed.
Time Frame: Day 28 and Day 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: NANOGRAM PER MILLILITER (NG/ML)
Arm/Group | CAMICINAL 25 MG | PLACEBO
Number analyzed (Participants) | 58 | 0
NANOGRAM PER MILLILITER (NG/ML)
  DAY 28: number analyzed (Participants) | 48 | 0
  DAY 28 | 171.746 (121.7083) |
  DAY 84: number analyzed (Participants) | 32 | 0
  DAY 84 | 166.382 (132.5696) |

ADVERSE EVENTS:
Time Frame: Up to end of follow up (100 days).
Description: Safety Population comprised of participants who received at least one dose of the study drug and were followed-up for at least one post-Baseline safety assessment; however, one participant randomized to Placebo arm had quantifiable concentration of camicinal in blood and therefore was analyzed in the camicinal group.
Arm/Group | CAMICINAL 25 MG | PLACEBO
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 3/58 | 2/56
Other Adverse Events (participants affected / at risk) | 22/58 | 27/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAMICINAL 25 MG (N=58) | PLACEBO (N=56)
VERTIGO (Ear and labyrinth disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 2 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAMICINAL 25 MG (N=58) | PLACEBO (N=56)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 3
DIARRHOEA (Gastrointestinal disorders) | 3 | 4
FLATULENCE (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 4
VOMITING (Gastrointestinal disorders) | 0 | 5
FATIGUE (General disorders) | 2 | 1
BRONCHITIS (Infections and infestations) | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
SINUSITIS (Infections and infestations) | 1 | 2
TOOTH INFECTION (Infections and infestations) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 4
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 2 | 0
HEADACHE (Nervous system disorders) | 4 | 7
DEPRESSION (Psychiatric disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.